CLINICAL TRIAL: NCT03404557
Title: Proteomic Analysis of Crohn's Disease Macrophages in Response or Not to Adherent-Invasive Escherichia Coli
Brief Title: Proteomic Analysis of Crohn's Disease Macrophages in Response or Not to AIEC
Acronym: ROMAN
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Laboratoire M2Ish (Unknown)
Responsible Party: Sponsor
Other Study IDs: CHU-370; 2017-A00667-46 (Other: 2017-A00667-46)
Record Dates: First submitted 2018-01-12; First posted 2018-01-19 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Crohn's Disease; Ulcerative Colitis
Keywords: Crohn's Disease; Ulcerative colitis; Macrophages; Adherent-Invasive Escherichia coli; Proteomic analysis
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Crohn's Disease patients group: 44 patients
  Interventions: Other: Proteomic analysis
- Ulcerative Colitis patients group: 22 patients
  Interventions: Other: Proteomic analysis
- Healthy volunteers group: 22 patients
  Interventions: Other: Proteomic analysis

INTERVENTIONS:
Other: Proteomic analysis — Proteomic analysis of Crohn's disease macrophages in response or not to Adherent-Invasive Escherichia coli

SUMMARY:
The M2iSH laboratory showed with two previous clinical trials that Crohn's Disease (CD) macrophages present i) a defect to control Adherent-Invasive Escherichia coli (AIEC) infection related to polymorphisms associated with CD; ii) a CD - specific cytokine secretion profile after an AIEC infection and intestinal inflammation dependent; iii) a modification of the response of CD macrophages at a basal state and after the AIEC infection. These results consolidate the hypothesis of a defect specific to CD macrophages.

That's why, the primary purpose of this study is to realize a proteomic analysis of macrophages of CD patients infected or not with AIEC and to compare them to Ulcerative Colitis (UC) patients and healthy volunteers.

DETAILED DESCRIPTION:
The macrophages characterization will be realized at a basal state and in response or not to AIEC.

Investigator aimed to 1) better understand the differences between macrophages of CD patients, UC patients and healthy volunteers but also the impact of AIEC infection on these macrophages to provide key informations to detect and characterize the defect of these macrophages; 2) highlight one or several protein in CD macrophages that could represent, in a long term, a potential therapeutic target of CD.

ELIGIBILITY:
Inclusion Criteria:

* - Crohn's Disease or ulcerative colitis or healthy volunteers
* Age > 18 years
* Patients benefiting from the health insurance plan
* Patients who can read and attest to understanding the information note and informed consent

Exclusion Criteria:

* Pregnant or breastfeeding woman
* Under guardianship or curatorship
* Refusing the genetic part of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Crohn's disease
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2018-01-18 (Actual); Primary Completion 2019-01-18 (Actual); Study Completion 2019-01-18 (Actual)

PRIMARY OUTCOMES:
Compare the proteomic profile of macrophages of patients with CD to patients with UC and healthy subjects in the basal state | at day 1
  Compare concentrations of different protein types in the supernatant of macrophages from patients with CD through proteomic approaches, compared with patients with UC or controls.

SECONDARY OUTCOMES:
Comparison of concentrations of different protein types in the supernatant of macrophages | at day 1
presence of subgroups of patients with CD based on the proteomic profile of their macrophages. | at day 1
association between these subgroups of patients with CD and biological parameters. | at day 1
associations between the proteomic profiles of macrophages of patients with CD, UC or control subjects and fecal AIEC status | at day 1
associations between the levels of entry, survival and multiplication of AIEC bacteria | at day 1
impact of anti-TNF treatment on the proteomic profile (s) observed for macrophages of patients with CD | at day 1
associations between the Proteomic profile (s) of the macrophages derived from monocytes and their AIEC status | at day 1
associations between the Proteomic profile (s) of tissue macrophages and their AIEC status | at day 1

CONTACTS AND LOCATIONS:
Overall Officials: Anthony BUISSON, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France